CLINICAL TRIAL: NCT02737579
Title: XFM: (X-ray Fused With MRI) Guided Cardiac Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joshua Kanter (Other)
Responsible Party: Sponsor-Investigator, Joshua Kanter, Joshua Kanter, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3879; Internal Bridge Funding (Other Grant/Funding Number: Children's Research Institute, Children's National)
Record Dates: First submitted 2016-02-17; First posted 2016-04-14 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Congenital Heart Defect
Keywords: cardiac catheterization; cardiac MRI
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XFM guidance (Other): X-ray fused cardiac MRI images used for guidance tool to perform cardiac catheterization procedure
  Interventions: Procedure: XFM guidance

INTERVENTIONS:
Procedure: XFM guidance — X-ray images and MRI roadmaps are aligned, during the medically indicated catheterization procedure, both conventional X-ray and investigational XFM images are displayed side-by-side. The operator may choose to be guided by either.

SUMMARY:
This study will evaluate the use of x-ray fused with MR images as an imaging tool to help guide catheter tools during diagnostic and therapeutic cardiac catheterization procedures.

DETAILED DESCRIPTION:
Cardiovascular interventional procedures are currently conducted under the guidance of X-ray fluoroscopy. Magnetic resonance imaging (MRI) can provide increased soft tissue information about the cardiovascular system. By combining the familiar X-ray environment with superior magnetic resonance imaging, the investigator hopes to enhance and expand the capabilities of cardiac catheterization techniques.

The investigator will conduct cardiac catheterization procedures using XFM guidance in pediatric research patients who are undergoing medically necessary procedures. The investigator aims to decrease the exposure of these patients to the routine hazards of ionizing radiation and contrast exposure compared to the standard of care approach.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adults of any age
2. Undergoing clinically-indicated cardiovascular catheterization

Exclusion Criteria:

1. Cardiovascular instability precluding baseline medially-necesary MRI
2. Women who are pregnant
3. Women who are nursing and who do not plan to discard breast milk for 24 hours
4. All patients who are medically judged to have contraindication(s) to MRI scanning. Contraindications include implanted metal devices which are contraindicated for MRI scanning

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-07-23 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Radiation exposure measurement | At the end of each catheterization procedure through study completion,up to 8 years.
  Comparisons with data from historical controls undergoing matched invasive cardiology procedures at Children's National Medical Center

SECONDARY OUTCOMES:
Fluoroscopy time measurement | At the end of each catheterization procedure through study completion,up to 8 years.
  Comparisons with data from historical controls undergoing matched procedures at Children's National Medical Center
Contrast volume measurement | At the end of each catheterization procedure through study completion, up to 8 years.
  Comparisons with data from historical controls undergoing matched invasive cardiology procedures at Children's National Medical Center will be examined.
Procedure time measurement | At the end of each catheterization procedure through study completion,up to 8 years.
  Comparisons with data from historical controls undergoing matched procedures at Children's National Medical Center

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Kanter, MD, Principal Investigator — Children's National Hospital System
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Silva R, Gutierrez LF, Raval AN, McVeigh ER, Ozturk C, Lederman RJ. X-ray fused with magnetic resonance imaging (XFM) to target endomyocardial injections: validation in a swine model of myocardial infarction. Circulation. 2006 Nov 28;114(22):2342-50. doi: 10.1161/CIRCULATIONAHA.105.598524. Epub 2006 Nov 13. PMID 17101858
- [Background] Gutierrez LF, Silva Rd, Ozturk C, Sonmez M, Stine AM, Raval AN, Raman VK, Sachdev V, Aviles RJ, Waclawiw MA, McVeigh ER, Lederman RJ. Technology preview: X-ray fused with magnetic resonance during invasive cardiovascular procedures. Catheter Cardiovasc Interv. 2007 Nov 15;70(6):773-82. doi: 10.1002/ccd.21352. PMID 18022851
- [Background] Faranesh AZ, Kellman P, Ratnayaka K, Lederman RJ. Integration of cardiac and respiratory motion into MRI roadmaps fused with x-ray. Med Phys. 2013 Mar;40(3):032302. doi: 10.1118/1.4789919. PMID 23464334
- [Background] George AK, Sonmez M, Lederman RJ, Faranesh AZ. Robust automatic rigid registration of MRI and X-ray using external fiducial markers for XFM-guided interventional procedures. Med Phys. 2011 Jan;38(1):125-41. doi: 10.1118/1.3523621. PMID 21361182
- [Background] Gutierrez LF, Ozturk C, McVeigh ER, Lederman RJ. A practical global distortion correction method for an image intensifier based x-ray fluoroscopy system. Med Phys. 2008 Mar;35(3):997-1007. doi: 10.1118/1.2839099. PMID 18404935
- [Background] Kleinerman RA. Cancer risks following diagnostic and therapeutic radiation exposure in children. Pediatr Radiol. 2006 Sep;36 Suppl 2(Suppl 2):121-5. doi: 10.1007/s00247-006-0191-5. PMID 16862418
- [Background] Andreassi MG, Ait-Ali L, Botto N, Manfredi S, Mottola G, Picano E. Cardiac catheterization and long-term chromosomal damage in children with congenital heart disease. Eur Heart J. 2006 Nov;27(22):2703-8. doi: 10.1093/eurheartj/ehl014. Epub 2006 May 22. PMID 16717079
- [Background] Beels L, Bacher K, De Wolf D, Werbrouck J, Thierens H. gamma-H2AX foci as a biomarker for patient X-ray exposure in pediatric cardiac catheterization: are we underestimating radiation risks? Circulation. 2009 Nov 10;120(19):1903-9. doi: 10.1161/CIRCULATIONAHA.109.880385. Epub 2009 Oct 26. PMID 19858412
- [Background] Schwartz GJ, Haycock GB, Edelmann CM Jr, Spitzer A. A simple estimate of glomerular filtration rate in children derived from body length and plasma creatinine. Pediatrics. 1976 Aug;58(2):259-63. PMID 951142
- [Background] Kiringoda R, Thurm AE, Hirschtritt ME, Koziol D, Wesley R, Swedo SE, O'Grady NP, Quezado ZM. Risks of propofol sedation/anesthesia for imaging studies in pediatric research: eight years of experience in a clinical research center. Arch Pediatr Adolesc Med. 2010 Jun;164(6):554-60. doi: 10.1001/archpediatrics.2010.75. PMID 20530306
- [Background] Haustein J, Laniado M, Niendorf HP, Louton T, Beck W, Planitzer J, Schoffel M, Reiser M, Kaiser W, Schorner W, et al. Triple-dose versus standard-dose gadopentetate dimeglumine: a randomized study in 199 patients. Radiology. 1993 Mar;186(3):855-60. doi: 10.1148/radiology.186.3.8430199.
- [Background] Niendorf HP, Alhassan A, Geens VR, Clauss W. Safety review of gadopentetate dimeglumine. Extended clinical experience after more than five million applications. Invest Radiol. 1994 Jun;29 Suppl 2:S179-82. doi: 10.1097/00004424-199406001-00059. No abstract available. PMID 7928222
- [Background] Niendorf HP, Dinger JC, Haustein J, Cornelius I, Alhassan A, Clauss W. Tolerance data of Gd-DTPA: a review. Eur J Radiol. 1991 Jul-Aug;13(1):15-20. doi: 10.1016/0720-048x(91)90049-2. PMID 1889423
- [Background] Niendorf HP, Haustein J, Cornelius I, Alhassan A, Clauss W. Safety of gadolinium-DTPA: extended clinical experience. Magn Reson Med. 1991 Dec;22(2):222-8; discussion 229-32. doi: 10.1002/mrm.1910220212. PMID 1812350
- [Background] Niendorf HP, Haustein J, Louton T, Beck W, Laniado M. Safety and tolerance after intravenous administration of 0.3 mmol/kg Gd-DTPA. Results of a randomized, controlled clinical trial. Invest Radiol. 1991 Nov;26 Suppl 1:S221-3; discussion S232-5. doi: 10.1097/00004424-199111001-00075. No abstract available. PMID 1808134
- [Background] Dillman JR, Ellis JH, Cohan RH, Strouse PJ, Jan SC. Frequency and severity of acute allergic-like reactions to gadolinium-containing i.v. contrast media in children and adults. AJR Am J Roentgenol. 2007 Dec;189(6):1533-8. doi: 10.2214/AJR.07.2554. PMID 18029897
- [Background] Sundgren PC, Leander P. Is administration of gadolinium-based contrast media to pregnant women and small children justified? J Magn Reson Imaging. 2011 Oct;34(4):750-7. doi: 10.1002/jmri.22413. PMID 21928308
- [Background] Deo A, Fogel M, Cowper SE. Nephrogenic systemic fibrosis: a population study examining the relationship of disease development to gadolinium exposure. Clin J Am Soc Nephrol. 2007 Mar;2(2):264-7. doi: 10.2215/CJN.03921106. Epub 2007 Feb 7. PMID 17699423